CLINICAL TRIAL: NCT03148080
Title: Work Ability in Young Adult Survivors (WAYS)
Brief Title: Work Ability in Young Adult Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00045363; NCI-2017-00991 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WF 10217 (Other: Wake Forest NCORP Research Base); WF-10217 (Other: DCP); WF-10217 (Other: CTEP); P30CA012197 (NIH); R21CA191989 (NIH); UG1CA189824 (NIH); NCI-2017-00991 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-05-05; First posted 2017-05-10 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Cancer Survivor
MeSH Terms: interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Participants complete a Current Medical Conditions Form, the CogState web-based cognitive assessment, and a Self-Report Questionnaire administration over 45-60 minutes containing measures of work ability and other work-related measures, cognitive, physical, and psychosocial symptoms, and characteristics of workplace environment. Self-report measures of individual and family characteristics, resources, and demands are also included.
  Interventions: Procedure: Cognitive Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Cognitive Assessment — Complete CogState
Other: Questionnaire Administration — Complete Self-Report Questionnaire

SUMMARY:
To document levels of labor force participation, occupation, educational attainment, and financial toxicity following cancer treatment in YA cancer survivors aged 25-34 years.

DETAILED DESCRIPTION:
This observational, cross-sectional study will recruit 220 analyzable YA survivors through the Wake Forest National Cancer Institute Community Oncology Research Program (NCORP) Research Base (WF NCORP RB). Data will be collected using a web-based interface and will capture physical, psychosocial and cognitive late effects; work ability; work-related outcomes, including labor force participation, occupation, work place characteristics, and educational attainment; survivor characteristics; and cancer diagnosis/treatment information (from clinical records). We will evaluate the relationships among these measures using the theoretical framework to guide statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* >= 2 to < 10 years post-cancer diagnosis (per diagnostic pathology report)
* Diagnosed with first cancer (any type except types listed in exclusion criteria below) at age >= 15 years
* Ability to understand and willingness to sign a written informed consent document
* Must be able to read and understand English

Exclusion Criteria:

* Currently receiving active cancer treatment (acceptable to be on maintenance or hormonal therapies)
* Life expectancy less than 6 months
* Precancerous or pre invasive conditions (myelodysplastic syndrome; carcinoma in situ; non-melanoma skin cancer) without progression to malignancy without another prior primary cancer diagnosis; (those who have had these conditions may participate IF they have a primary cancer diagnosis)
* Non-Hispanic Whites (effective 11/01/2018)

Ages: 25 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Currently Employed | Baseline
  Labor force participation will be summarized as employed, unemployed (not working, but looking for work), and not in labor force (not employed and not looking for work or active duty military).
Occupation Status | Baseline
  This categorical work-related outcomes will be described using frequencies. Occupational status will be summarized using the 2010 Standard Occupational Classification (SOC) system: managerial and professional) (SOC major groups 11-29), (support, retail, and service (SOC major groups 31-43), and construction, production and transportation (SOC major groups 45-53).
Educational Attainment | Baseline
  This categorical work-related outcomes will be described using frequencies. Educational attainment will be classified as using the Current Population Survey classifications so that we can compare rates to US Benchmarks. The classifications are the following: Less than 1st grade, 1-4th grade, 5th-6th grade, 7-8th grade, 9th grade, 10th grade, 11th grade, 12 grade (no diploma), high school diploma or equivalent, some college (no degree), associate degree in college - occupational/vocational program, associate degree in college - academic program, Bachelor's degree, Master's degree, Professional School Degree (MD, DDS, DVM, JD etc.), Doctorate Degree.
Financial Toxicity | Baseline
  The Comprehensive Score for Financial Toxicity (COST) is a self-report measure of financial distress experienced in response to cancer and its treatment. It ranges from 0-44, with higher scores associated with greater financial toxicity.

SECONDARY OUTCOMES:
Work ability (measured by Work Ability Index global score) | Baseline
  The Work Ability Index score ranges from 7 to 49, with higher scores indicating better workability; the Work Ability Index (WAI) global score is an item within the Work Ability Index which measures work ability from 0 to 10, with 10 representing the best work ability.
Work ability (measured by Work Ability Index) | Baseline
  The Work Ability Index (WAI) score ranges from 7 to 49, with higher scores indicating better workability; the Work Ability Index (WAI) global score is an item within the Work Ability Index which measures work ability from 0 to 10, with 10 representing the best work ability.
Work ability measured by Work Limitations Questionnaire score | Baseline
  The Work Limitations Questionnaire (WLQ) is a self-report measure of impact of chronic health conditions/treatment on job performance. Subscales: (1) time demands; (2) physical demands; (3) mental-interpersonal demands; and (4) output demands. Scale scores range from 0 (limited none of the time) to 100 (limited all of the time) with 0 being better.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Danhauer, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (327):
- United States (326):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - McKee Medical Center, Loveland, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Blank Children's Hospital, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - JCHC McCreery Cancer Center, Fairfield, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Bronson Battle Creek, Battle Creek, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Spartanburg Medical Center - Mary Black Campus, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Sovah Health Martinsville, Martinsville, Virginia
  - Jefferson Healthcare, Port Townsend, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
- FHP Health Center-Guam, Tamuning, Guam

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration.
Access Criteria: upon request to NCORP@wakehealth.edu

REFERENCES:
- [Background] Feuerstein M, Harrington CB. Recommendations for the U.S. National Occupational Research Agenda: research on cancer survivorship and musculoskeletal disorders and work disability. J Occup Rehabil. 2006 Mar;16(1):1-5. doi: 10.1007/s10926-005-9004-1. PMID 16688488
- [Background] Patrick DL, Ferketich SL, Frame PS, Harris JJ, Hendricks CB, Levin B, Link MP, Lustig C, McLaughlin J, Ried LD, Turrisi AT 3rd, Unutzer J, Vernon SW; National Institutes of Health State-of-the-Science Panel. National Institutes of Health State-of-the-Science Conference Statement: Symptom Management in Cancer: Pain, Depression, and Fatigue, July 15-17, 2002. J Natl Cancer Inst. 2003 Aug 6;95(15):1110-7. doi: 10.1093/jnci/djg014. PMID 12902440
- [Background] The President's Cancer Panel. Living Beyond Cancer: Finding New Balance, President's Cancer Panel 2003-2004 Annual Report. U.S. Department of Health and Human Services, National Institutes of Health.; 2004
- [Background] Munir F, Yarker J, McDermott H. Employment and the common cancers: correlates of work ability during or following cancer treatment. Occup Med (Lond). 2009 Sep;59(6):381-9. doi: 10.1093/occmed/kqp088. PMID 19692524
- [Background] Closing the Gap: A Strategic Plan Addressing the Recommendations of the Adolescent and Young Adult Oncology Progress Review Group. National Institutes of Health; 2007
- [Background] Bellizzi KM, Smith A, Schmidt S, Keegan TH, Zebrack B, Lynch CF, Deapen D, Shnorhavorian M, Tompkins BJ, Simon M; Adolescent and Young Adult Health Outcomes and Patient Experience (AYA HOPE) Study Collaborative Group. Positive and negative psychosocial impact of being diagnosed with cancer as an adolescent or young adult. Cancer. 2012 Oct 15;118(20):5155-62. doi: 10.1002/cncr.27512. Epub 2012 Mar 13. PMID 22415815
- [Background] Keegan TH, Lichtensztajn DY, Kato I, Kent EE, Wu XC, West MM, Hamilton AS, Zebrack B, Bellizzi KM, Smith AW; AYA HOPE Study Collaborative Group. Unmet adolescent and young adult cancer survivors information and service needs: a population-based cancer registry study. J Cancer Surviv. 2012 Sep;6(3):239-50. doi: 10.1007/s11764-012-0219-9. Epub 2012 Mar 29. PMID 22457219
- [Background] Tai E, Buchanan N, Townsend J, Fairley T, Moore A, Richardson LC. Health status of adolescent and young adult cancer survivors. Cancer. 2012 Oct 1;118(19):4884-91. doi: 10.1002/cncr.27445. Epub 2012 Jun 11. PMID 22688896
- [Background] Kirchhoff AC, Lyles CR, Fluchel M, Wright J, Leisenring W. Limitations in health care access and utilization among long-term survivors of adolescent and young adult cancer. Cancer. 2012 Dec 1;118(23):5964-72. doi: 10.1002/cncr.27537. Epub 2012 Sep 24. PMID 23007632
- [Background] de Boer AG, Frings-Dresen MH. Employment and the common cancers: return to work of cancer survivors. Occup Med (Lond). 2009 Sep;59(6):378-80. doi: 10.1093/occmed/kqp087. PMID 19692523
- [Background] Taskila T, Martikainen R, Hietanen P, Lindbohm ML. Comparative study of work ability between cancer survivors and their referents. Eur J Cancer. 2007 Mar;43(5):914-20. doi: 10.1016/j.ejca.2007.01.012. Epub 2007 Feb 20. PMID 17314041
- [Background] Moran JR, Short PF, Hollenbeak CS. Long-term employment effects of surviving cancer. J Health Econ. 2011 May;30(3):505-14. doi: 10.1016/j.jhealeco.2011.02.001. Epub 2011 Mar 1. PMID 21429606
- [Background] Hansen JA, Feuerstein M, Calvio LC, Olsen CH. Breast cancer survivors at work. J Occup Environ Med. 2008 Jul;50(7):777-84. doi: 10.1097/JOM.0b013e318165159e. PMID 18617833
- [Background] Oberst K, Bradley CJ, Gardiner JC, Schenk M, Given CW. Work task disability in employed breast and prostate cancer patients. J Cancer Surviv. 2010 Dec;4(4):322-30. doi: 10.1007/s11764-010-0128-8. Epub 2010 Jun 12. PMID 20549572
- [Background] Short PF, Vasey JJ, Tunceli K. Employment pathways in a large cohort of adult cancer survivors. Cancer. 2005 Mar 15;103(6):1292-301. doi: 10.1002/cncr.20912. PMID 15700265
- [Background] Taskila T, Lindbohm ML. Factors affecting cancer survivors' employment and work ability. Acta Oncol. 2007;46(4):446-51. doi: 10.1080/02841860701355048. PMID 17497311
- [Background] Parsons HM, Harlan LC, Lynch CF, Hamilton AS, Wu XC, Kato I, Schwartz SM, Smith AW, Keel G, Keegan TH. Impact of cancer on work and education among adolescent and young adult cancer survivors. J Clin Oncol. 2012 Jul 1;30(19):2393-400. doi: 10.1200/JCO.2011.39.6333. Epub 2012 May 21. PMID 22614977
- [Background] LIVESTRONG Report Committee. "I Learned to Live with It" is Not Good Enough: Challenges Reported by Post-Treatment Cancer Survivors in the LIVESTRONG Surveys: A LIVESTRONG Report, 2010. Lance Armstrong Foundation; 2010. _http://livestrong.org/_. Accessed January 28, 2013
- [Background] Kirchhoff AC, Krull KR, Ness KK, Armstrong GT, Park ER, Stovall M, Robison LL, Leisenring W. Physical, mental, and neurocognitive status and employment outcomes in the childhood cancer survivor study cohort. Cancer Epidemiol Biomarkers Prev. 2011 Sep;20(9):1838-49. doi: 10.1158/1055-9965.EPI-11-0239. Epub 2011 Aug 15. PMID 21844244
- [Background] Ness KK, Gurney JG, Zeltzer LK, Leisenring W, Mulrooney DA, Nathan PC, Robison LL, Mertens AC. The impact of limitations in physical, executive, and emotional function on health-related quality of life among adult survivors of childhood cancer: a report from the Childhood Cancer Survivor Study. Arch Phys Med Rehabil. 2008 Jan;89(1):128-36. doi: 10.1016/j.apmr.2007.08.123. PMID 18164342
- [Background] Ness KK, Hudson MM, Ginsberg JP, Nagarajan R, Kaste SC, Marina N, Whitton J, Robison LL, Gurney JG. Physical performance limitations in the Childhood Cancer Survivor Study cohort. J Clin Oncol. 2009 May 10;27(14):2382-9. doi: 10.1200/JCO.2008.21.1482. Epub 2009 Mar 30. PMID 19332713
- [Background] Kirchhoff AC, Krull KR, Ness KK, Park ER, Oeffinger KC, Hudson MM, Stovall M, Robison LL, Wickizer T, Leisenring W. Occupational outcomes of adult childhood cancer survivors: A report from the childhood cancer survivor study. Cancer. 2011 Jul 1;117(13):3033-44. doi: 10.1002/cncr.25867. Epub 2011 Jan 18. PMID 21246530
- [Background] Kirchhoff AC, Leisenring W, Krull KR, Ness KK, Friedman DL, Armstrong GT, Stovall M, Park ER, Oeffinger KC, Hudson MM, Robison LL, Wickizer T. Unemployment among adult survivors of childhood cancer: a report from the childhood cancer survivor study. Med Care. 2010 Nov;48(11):1015-25. doi: 10.1097/MLR.0b013e3181eaf880. PMID 20940653
- [Background] Haas SA, Fosse NE. Health and the educational attainment of adolescents: evidence from the NLSY97. J Health Soc Behav. 2008 Jun;49(2):178-92. doi: 10.1177/002214650804900205. PMID 18649501
- [Background] Jackson MI. Understanding links between adolescent health and educational attainment. Demography. 2009 Nov;46(4):671-94. doi: 10.1353/dem.0.0078. PMID 20084824
- [Background] Haas SA. Health selection and the process of social stratification: the effect of childhood health on socioeconomic attainment. J Health Soc Behav. 2006 Dec;47(4):339-54. doi: 10.1177/002214650604700403. PMID 17240924
- [Background] Case A, Fertig A, Paxson C. The lasting impact of childhood health and circumstance. J Health Econ. 2005 Mar;24(2):365-89. doi: 10.1016/j.jhealeco.2004.09.008. Epub 2005 Jan 5. PMID 15721050
- [Background] Feuerstein M, Todd BL, Moskowitz MC, Bruns GL, Stoler MR, Nassif T, Yu X. Work in cancer survivors: a model for practice and research. J Cancer Surviv. 2010 Dec;4(4):415-37. doi: 10.1007/s11764-010-0154-6. Epub 2010 Oct 14. PMID 20945110
- [Background] Behling O, Law KS. Translating Questionnaires and Other Research Insturments: Problems and Solutions. Sage paper series; 2000
- [Background] WAI Online Questionnaire (Short Version) WAI Netzwerk. Bergische Universitat Wuppertal.; 2013
- [Background] Tuomi K., Ilmarinen J, Katajarinne L, A. T. Work Ability Index. 2nd revised. Helsinki: Finnish Institute of Occupational Health, 1998; 1998
- [Background] Lindbohm ML, Taskila T, Kuosma E, Hietanen P, Carlsen K, Gudbergsson S, Gunnarsdottir H. Work ability of survivors of breast, prostate, and testicular cancer in Nordic countries: a NOCWO study. J Cancer Surviv. 2012 Mar;6(1):72-81. doi: 10.1007/s11764-011-0200-z. Epub 2011 Nov 2. PMID 22042662
- [Background] de Boer AG, Verbeek JH, Spelten ER, Uitterhoeve AL, Ansink AC, de Reijke TM, Kammeijer M, Sprangers MA, van Dijk FJ. Work ability and return-to-work in cancer patients. Br J Cancer. 2008 Apr 22;98(8):1342-7. doi: 10.1038/sj.bjc.6604302. Epub 2008 Mar 18. PMID 18349834
- [Background] Lerner D, Amick BC 3rd, Rogers WH, Malspeis S, Bungay K, Cynn D. The Work Limitations Questionnaire. Med Care. 2001 Jan;39(1):72-85. doi: 10.1097/00005650-200101000-00009. PMID 11176545
- [Background] Calvio L, Peugeot M, Bruns GL, Todd BL, Feuerstein M. Measures of cognitive function and work in occupationally active breast cancer survivors. J Occup Environ Med. 2010 Feb;52(2):219-27. doi: 10.1097/JOM.0b013e3181d0bef7. PMID 20134340
- [Background] Feuerstein M, Hansen JA, Calvio LC, Johnson L, Ronquillo JG. Work productivity in brain tumor survivors. J Occup Environ Med. 2007 Jul;49(7):803-11. doi: 10.1097/JOM.0b013e318095a458. PMID 17622854
- [Background] Smith TW, Marsden PV, Michael H, Jiburm K. General Social Surveys, 1972-2012: Cumulative Codebook / Principal Investigator, Tom W. Smith; Co-Principal Investigators, Peter V. Marsden and Michael Hout. 2nd revised. -- Chicago: National Opinion Research Center, 2013. 3,422 pp.,: National Data Program for the Social Sciences Series, no. 21; 2013.
- [Background] Standard Occupational Classification Committee (SOCPC) 2010 SOC Definitions. U.S. Bureau of Labor Statistics. (Updated January 2013) 2010 SOC User Guide.U.S.Bureau of Labor Statistics _www.bls.gov/soc/soc_2010_definitions.pdf_; 2010
- [Background] Gershon RC. Need for Cognitive Measures. In: National Institute on Disability and Rehabilitation. ; 2012.
- [Background] Maruff P, Thomas E, Cysique L, Brew B, Collie A, Snyder P, Pietrzak RH. Validity of the CogState brief battery: relationship to standardized tests and sensitivity to cognitive impairment in mild traumatic brain injury, schizophrenia, and AIDS dementia complex. Arch Clin Neuropsychol. 2009 Mar;24(2):165-78. doi: 10.1093/arclin/acp010. Epub 2009 Mar 25. PMID 19395350
- [Background] Phillips KM, Jim HS, Donovan KA, Pinder-Schenck MC, Jacobsen PB. Characteristics and correlates of sleep disturbances in cancer patients. Support Care Cancer. 2012 Feb;20(2):357-65. doi: 10.1007/s00520-011-1106-z. Epub 2011 Feb 11. PMID 21311913
- [Background] Hinchcliff M, Beaumont JL, Thavarajah K, Varga J, Chung A, Podlusky S, Carns M, Chang RW, Cella D. Validity of two new patient-reported outcome measures in systemic sclerosis: Patient-Reported Outcomes Measurement Information System 29-item Health Profile and Functional Assessment of Chronic Illness Therapy-Dyspnea short form. Arthritis Care Res (Hoboken). 2011 Nov;63(11):1620-8. doi: 10.1002/acr.20591. PMID 22034123
- [Background] Garcia SF, Cella D, Clauser SB, Flynn KE, Lad T, Lai JS, Reeve BB, Smith AW, Stone AA, Weinfurt K. Standardizing patient-reported outcomes assessment in cancer clinical trials: a patient-reported outcomes measurement information system initiative. J Clin Oncol. 2007 Nov 10;25(32):5106-12. doi: 10.1200/JCO.2007.12.2341. PMID 17991929
- [Background] Jensen RE, Potosky AL, Reeve BB, Hahn E, Cella D, Fries J, Smith AW, Keegan TH, Wu XC, Paddock L, Moinpour CM. Validation of the PROMIS physical function measures in a diverse US population-based cohort of cancer patients. Qual Life Res. 2015 Oct;24(10):2333-44. doi: 10.1007/s11136-015-0992-9. Epub 2015 May 3. PMID 25935353
- [Background] Wagner LI, Schink J, Bass M, Patel S, Diaz MV, Rothrock N, Pearman T, Gershon R, Penedo FJ, Rosen S, Cella D. Bringing PROMIS to practice: brief and precise symptom screening in ambulatory cancer care. Cancer. 2015 Mar 15;121(6):927-34. doi: 10.1002/cncr.29104. Epub 2014 Nov 6. PMID 25376427
- [Background] de Souza JA, Yap BJ, Hlubocky FJ, Wroblewski K, Ratain MJ, Cella D, Daugherty CK. The development of a financial toxicity patient-reported outcome in cancer: The COST measure. Cancer. 2014 Oct 15;120(20):3245-53. doi: 10.1002/cncr.28814. Epub 2014 Jun 20. PMID 24954526
- [Background] Salsman JM, Lai JS, Hendrie HC, Butt Z, Zill N, Pilkonis PA, Peterson C, Stoney CM, Brouwers P, Cella D. Assessing psychological well-being: self-report instruments for the NIH Toolbox. Qual Life Res. 2014 Feb;23(1):205-15. doi: 10.1007/s11136-013-0452-3. Epub 2013 Jun 16. PMID 23771709
- [Background] Diener E, Wirtz D, Tov W, Kim-Prieto C, Choi D, Oishi S, Biswas-Diener R. New measures of well-being: Flourishing and positive and negative feelings. Soc Indic Res. 2010;39:247-266.
- [Background] Cann A, Calhoun LG, Tedeschi RG, Taku K, Vishnevsky T, Triplett KN, Danhauer SC. A short form of the Posttraumatic Growth Inventory. Anxiety Stress Coping. 2010;23(2):127-37. doi: 10.1080/10615800903094273. PMID 19582640
- [Background] Lindbohm ML, Kuosma E, Taskila T, Hietanen P, Carlsen K, Gudbergsson S, Gunnarsdottir H. Cancer as the cause of changes in work situation (a NOCWO study). Psychooncology. 2011 Aug;20(8):805-12. doi: 10.1002/pon.1797. Epub 2010 Jul 11. PMID 20623820
- [Background] Torp S, Nielsen RA, Gudbergsson SB, Dahl AA. Worksite adjustments and work ability among employed cancer survivors. Support Care Cancer. 2012 Sep;20(9):2149-56. doi: 10.1007/s00520-011-1325-3. Epub 2011 Nov 16. PMID 22086407
- [Background] Baker F, Denniston M, Smith T, West MM. Adult cancer survivors: how are they faring? Cancer. 2005 Dec 1;104(11 Suppl):2565-76. doi: 10.1002/cncr.21488. PMID 16258929
- [Background] Baker F, Denniston M, Zabora JR, Marcellus D. Cancer Problems in Living and Quality of Life After Bone Marrow Transplation. J Clin Psychol Med Settings. 2003;10(1):27-34. doi:10.1023/A:1022801713046.
- [Background] Zhao L, Portier K, Stein K, Baker F, Smith T. Exploratory factor analysis of the Cancer Problems in Living Scale: a report from the American Cancer Society's Studies of Cancer Survivors. J Pain Symptom Manage. 2009 Apr;37(4):676-86. doi: 10.1016/j.jpainsymman.2008.04.011. Epub 2008 Sep 11. PMID 18789641
- [Background] Lai JS, Butt Z, Wagner L, Sweet JJ, Beaumont JL, Vardy J, Jacobsen PB, Shapiro PJ, Jacobs SR, Cella D. Evaluating the dimensionality of perceived cognitive function. J Pain Symptom Manage. 2009 Jun;37(6):982-95. doi: 10.1016/j.jpainsymman.2008.07.012. PMID 19500722
- [Background] Beels CC, Gutwirth L, Berkeley J, Struening E. Measurements of social support in schizophrenia. Schizophr Bull. 1984;10(3):399-411. doi: 10.1093/schbul/10.3.399. PMID 6382589
- [Background] Brekke JS, Long JD, Kay DD. The structure and invariance of a model of social functioning in schizophrenia. J Nerv Ment Dis. 2002 Feb;190(2):63-72. doi: 10.1097/00005053-200202000-00001. PMID 11889358
- See also: Adolescent and Young Adult Cancer by Site: Incidence, Survival, and Mortality. National Cancer Institute Surveillance, Epidemiology, and End Results Program — http://seer.cancer.gov/archive/csr/1975_2011/results_merged/sect_32_aya.pdf
- See also: Bureau UC. Current Population Survey (CPS) — http://census.gov/programs-surveys/cps.html
- See also: Bureau UC. American Community Survey (ACS) — http://census.gov/programs-surveys/acs
- See also: HRS :: Documentation :: Questionnaires — http://hrsonline.isr.umich.edu/index.php?p=qnaires